CLINICAL TRIAL: NCT03090113
Title: A Random, Double-blind, Parallel, Placebo-controlled, Multi-center Study of Shuxuetong for Prevention of Recurrence in Acute Cerebrovascular Events With Embolism
Brief Title: Shuxuetong for Prevention of Recurrence in Acute Cerebrovascular Events With Embolism
Acronym: SPACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014ZX09201022-010-11
Record Dates: First submitted 2017-03-09; First posted 2017-03-24 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Embolic Stroke
Keywords: Stroke; Embolic Stroke; Shuxuetong; Recurrence; Symptomatic New Cerebral Infarction; Asymptomatic New Cerebral Infarction
MeSH Terms: conditions — Embolic Stroke; Stroke; Recurrence | interventions — shuxuetong

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shuxuetong Injection (Experimental): Shuxuetong Injection,12ml,ivgtt,day1; Shuxuetong Injection,6ml,ivgtt,day2 to day10;
  Interventions: Drug: Shuxuetong Injection
- Placebo Injection (Placebo Comparator): Placebo Injection,12ml,ivgtt,day1; Placebo Injection,6ml,ivgtt,day2 to day10;
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: Shuxuetong Injection — intravenous drip
  Other Names: Shuxuetong
  Arms: Shuxuetong Injection
Drug: Placebo Injection — intravenous drip
  Other Names: Placebo
  Arms: Placebo Injection

SUMMARY:
This is a randomized, double blind, placebo-controlled, parallel, multicenter research in order to evaluate the effect of Shuxuetong injection in prevention of symptomatic or asymptomatic new cerebral infarction within 10 days.

Subgroup study：Evaluate the role of advanced diagnostic technique in identifying potential causes of Embolic Stroke of Undetermined Source (ESUS).

DETAILED DESCRIPTION:
Shuxuetong injection or Placebo injection for 10days. About 2416 patients randomized at 80 centers all over China with 20 subgroup study centers.

Face to face interview at baseline, 10 days, and 90 days.

ELIGIBILITY:
Inclusion criteria

1. More than or equal to 18 years old and less than 80 years old;
2. Acute ischemic stroke, brain magnetic resonance imaging showed non lacunar infarction (subcortical infarction less than or equal to 1.5 cm);
3. Onset within 72 hours;
4. Patients or their family members are willing to sign the informed consent.

Exclusion criteria

1. Intracranial hemorrhage: cerebral hemorrhage, subarachnoid hemorrhage, etc.;
2. Transient ischemic attack;
3. Lacunar infarction;
4. History of acute stroke within 6 months;
5. Clear diagnosis of other causes of ischemic stroke (arterial dissection, arteritis, vasospasm, etc.);
6. The acute infarcts lesion more than one-half lobe in size;
7. Preceding modified Rankin Scale (mRS) score ≥ 2;
8. Cumulative usage of traditional Chinese medicine which activating blood circulation more than 3 times after onset, including but not limited to: Danhong, Xueshuantong, Xuesaitong, Ginkgo biloba, sodium ozagrel, Salvia miltiorrhiza, ligustrazine, Erigeron breviscapus, etc;
9. Chronic liver disease, liver and kidney dysfunction, lifted alanine aminotransferase (>3 times the ULN), lifted serum creatinine (>2 times the ULN）;
10. History of coagulopathy, systemic bleeding, thrombocytopenia or neutropenia;
11. Blood pressure >90/60 mmHg or ≤220/120 mmHg after treatment;
12. Serious heart or lung disease, in the judgment of clinical study staff, would not suitable to participant in the trial;
13. Patients with atrial fibrillation who were scheduled or likely to receive anticoagulant therapy with unfractionated heparin or low molecular weight heparin within 2 weeks after randomization
14. A medical condition likely to limit survival to less than three months or any other condition judged by the clinic team to likely limit the adherence to study procedures;
15. Known allergies for ingredients of the drug, allergy history for food or drug;
16. Pregnant, currently trying to become pregnant, or of child-bearing potential and not using birth control;
17. Participation in another clinical trial within 30 days;
18. Unable to understand and/or comply with the study procedures and/or follow-up studies due to mental illness, cognitive or emotional disorders.

Subgroup Exclusion Criteria

1. History of atrial fibrillation
2. Atrial fibrillation in 12-lead electrocardiogram (ECG);
3. Heart rate monitoring (dynamic electrocardiogram telemetry) up to 20 hours or more detected atrial fibrillation for 6 minutes or more;
4. Intracardiac thrombosis in thoracic or esophageal echocardiography;
5. Occlusion or proximal vessel infarction for more than 50%.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2416 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Symptomatic or Asymptomatic New Cerebral Infarction | 10 days
  Those patients who are still alive at 10 days after randomization will be contacted to set up a follow-up clinical visit. Information of recurrent symptomatic cerebral infarction will be collected and MRI examination will be performed to detect asymptomatic new cerebral infarction.

SECONDARY OUTCOMES:
Symptomatic Cerebral Infarction | 10 days
  Those patients who are still alive at 10 days after randomization will be contacted to set up a follow-up clinical visit. Information of recurrent symptomatic cerebral infarction will be collected.
Asymptomatic Cerebral Infarction | 10 days
  Those patients who are still alive at 10 days after randomization will be contacted to set up a follow-up clinical visit. MRI examination including diffusion weighted imaging (DWI) sequence will be performed.
Cerebral Infarction Volume Expansion | 10 days
  Those patients who are still alive at hospital discharge will be contacted to set up a follow-up clinical visit. MRI examination will be performed.
NIHSS Score Increase | 10 days
  Those patients who are still alive at hospital discharge will be contacted to set up a follow-up clinical visit. Neurological and functional assessments including NIHSS will be performed.
Recurrent Symptomatic Stroke(Cerebral infarction, cerebral hemorrhage) | 90 days
  Those patients who are still alive at 90days after onset will be contacted by telephone to set up a follow-up clinical visit. Information of recurrent symptomatic stroke will be collected.
Recurrent Symptomatic Ischemic Stroke | 90 days
  Those patients who are still alive at 90days after onset will be contacted by telephone to set up a follow-up clinical visit. Information of recurrent symptomatic ischmemic stroke will be collected.
Combined Vascular Events | 90 days
  Combined Vascular Events was defined as a combination of symptomatic stroke, myocardial infarction and vascular death.
Disability or Death | 90 days
  Disability or Death was defined as a score of 3 to 6 on the modified Rankin Scale at 90days after onset.

OTHER OUTCOMES:
Detected an Atrial Fibrillation Persistent ≥ 30s | 90 days
  Pre-specified Outcomes for Substudy of 'Etiology Study in Patients with ESUS'

CONTACTS AND LOCATIONS:
Overall Officials: Wang yongjun, MD, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
Locations (48):
- China (48):
  - Wuhu No.1 People's Hospital, Wuhu, Anhui
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Ansteel Group Hospital, Beijing, Beijing Municipality
  - Beiujing Fengtai Youanmen Hospital, Beijing, Beijing Municipality
  - The First Hospital of Fangshan District, Beijing, Beijing Municipality
  - Yongchuan hospital of Traditional Chinese Medicine, Chongqing, Chongqing Municipality
  - Houjie Hospital, Dongguan, Guangzhou
  - Cangzhou Peoole's Hospital, Cangzhou, Hebei
  - People's Hospital of Hejian, Cangzhou, Hebei
  - Kuancheng County Hospital, Chengde, Hebei
  - Traditional Chinese Medicine Hospital of Qiu County, Handan, Hebei
  - Hengshui Fourth Hospital, Hengshui, Hebei
  - Jizhou District Hospital of Hengshui, Hengshui, Hebei
  - Shijiazhuang Pingan Hospital Affiliated to Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - Heilongjiang Province Agricultural Reclamation Mudanjiang Authority Central Hospital, Mudanjiang, Heilongjiang
  - Handan Municipal Center Hospital, Handan, Henan
  - The First Affiliated Hospital of University of South China, Hengyang, Henan
  - People's Hospital of Zhongmu, Zhengzhou, Henan
  - Zhengzhou Yihe Hospital Affiliated to Henan University, Zhengzhou, Henan
  - Jingmen City Hospital of Traditional Chinese Medicine, Jingmen, Hubei
  - Wuhan NO.1 Hospital,Wuhan Hospital Of Traditional Chinese And Western Medicine, Wuhan, Hubei
  - Jiangsu Province Hospital of TCM, Nanjing, Jiangsu
  - Nantong 3rd People's Hospital, Nantong, Jiangsu
  - Zhangjiagang First People's Hospital, Suzhou, Jiangsu
  - Zhangjiagang Hospital of Traditional Chinese Medicine affiliated to Nanjing University of Chinese Medicine, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University-the Eastern Division, Changchun, Jilin
  - The Second People's Hospital of Huludao, Huludao, Liaoning
  - Jinzhou Medical University, Jinzhou, Liaoning
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Neimenggu
  - Wu Yuan People's Hospital, Bayan Nur, Neimenggu
  - Affiliated Hospital of Chifeng University, Chifeng, Neimenggu
  - Huimin People's Hospital, Binzhou, Shandong
  - People's Hospital of Penglai, Dengzhou, Shandong
  - Ningjin County People's Hospital, Dezhou, Shandong
  - Shandong Provincial Western Hospital, Jinan, Shandong
  - People's Hospital of Qingdao West Coast New Area, Qingdao, Shandong
  - Qingdao Haci medical group hospital, Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second People's Hospital of Shenzhen, Shenzhen, Shenzhen
  - Dongyang People's Hopital, Dongyang, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - No.1 People's Hospital of Taizhou, Taizhou, Zhejiang
  - Ruian People's Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gu HQ, Xie XW, Jing J, Meng X, Lv W, Yu JD, Lv XP, Li H, Wang YL, Wang YJ. Shuxuetong for Prevention of recurrence in Acute Cerebrovascular events with Embolism (SPACE) trial: rationale and design. Stroke Vasc Neurol. 2020 Sep;5(3):311-314. doi: 10.1136/svn-2019-000293. Epub 2020 Feb 27. PMID 32994371